CLINICAL TRIAL: NCT01236183
Title: Evaluation of Learning Curve of Manual Skills in Anesthesia Residents
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, kasana raksamani, Assoc Prof, Mahidol University
Other Study IDs: Si246/2553(E)
Record Dates: First submitted 2010-11-04; First posted 2010-11-08 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Intubation Skill; Laryngeal Mask Airway Insertion Skill; Spinal Anesthesia Skill; Epidural Anesthesia Skill; Radial Artery Cannulation Skill; Internal Jugular Vein Cannulation Skill
Keywords: manual skill; anesthesia residents

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine number of cases need to perform in new anesthesia residents to be proficient in manual skills.

DETAILED DESCRIPTION:
Manual skills in anesthesia are complex and unique to learn. The adequate cases need to be done to reach optimal success rate for each procedure is still varied from data available from the publications.

This study is designed to evaluate the number of cases need to perform in new anesthesia residents to be proficient in anesthesia skills, which are intubation, laryngeal mask insertion, spinal anesthesia, epidural anesthesia, radial artery cannulation and internal jugular vein cannulation.

ELIGIBILITY:
Inclusion Criteria:

* new anesthesia residents

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: new anesthesia residents
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kasana Raksamani, MD, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Bangkok, Thailand